CLINICAL TRIAL: NCT04615728
Title: APPENDICITIS DURING THE COVID-19 PANDEMIC: TO OPERATE OR NOT TO OPERATE, THAT IS THE QUESTION: COHORT STUDY FROM A TERTIARY CENTRE
Brief Title: MANAGEMENT OF APPENDICITIS DURING THE COVID-19 PANDEMIC
Acronym: observational
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: R Antakia, A Xanthis, F Georgiades, V Hudson, J Ashcroft, S Rooney, AA Singh, JR O'Neill, N Fearnhead, RH Hardwick, RJ Davies, John M Bennett (Unknown)
Responsible Party: Principal Investigator, Mr Ramez Antakia, Mr, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: PRN8996
Record Dates: First submitted 2020-11-02; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Acute Appendicitis
Keywords: acute appendicitis; COVID-19; conservative management; antibiotic therapy; laparoscopic appendicectomy; open surgery
MeSH Terms: conditions — Appendicitis; COVID-19 | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-COVID cohort: Patients recruited from 1st November 2019 to 9th March 2020
  Interventions: Procedure: laparoscopic or open appendicectomy
- COVID cohort: Patients recruited from 10th March 2020 to 5th July 2020
  Interventions: Procedure: laparoscopic or open appendicectomy

INTERVENTIONS:
Procedure: laparoscopic or open appendicectomy — Laparoscopic/open appendicectomy versus conservative management with antibiotic therapy with or without image-guided drainage of appendicular abscess/collection
  Other Names: conservative antibiotic therapy

SUMMARY:
During the Covid-19 pandemic, non-operative management for acute appendicitis (AA) was implemented in the UK. The aim of this study was to determine the efficacy and outcomes of conservative versus surgical management of AA during the pandemic.

DETAILED DESCRIPTION:
This prospective observational cohort study was conducted in a single UK tertiary referral centre and was registered locally as a clinical audit. Patients included in this study were adults (≥16 years) with a diagnosis of acute appendicitis made clinically and/or radiologically in our hospital. Patients presented sequentially to the emergency department, and subsequently were referred to the emergency surgical service for further management. The data collection periods were between 1st November 2019 and 10th March 2020 ('the pre-COVID period') and 10th March 2020 to 5th July 2020 ('COVID period'). The start of the COVID period was determined as the day of our hospital pandemic policy introduction, following the identification of the first SARS-CoV-2 positive patient at our site.

Data were collected retrospectively for the pre-COVID period and prospectively during the COVID pandemic using the electronic patient record (HYPERSPACE® Epic 2014 Version IU1, Epic Systems Corporation, Verona, WI, USA). Data collected included patient demographics, radiology reports, timings of consultations, operative records, post-operative care, post-operative complications, re-operation rate, length of hospital stay (LOS), histology results, re-attendance to hospital and mortality within 90 days of the initial presentation.

Study participants were scored using the Alvarado score (9), Appendicitis inflammatory response (AIR) score (10), the Adult appendicitis score (AAS) (11), American Society of Anaesthesiologists (ASA) physical status classification (12) and Rockwood Clinical Frailty Scale (13) based on their initial presentation history and investigations, as previously described in the literature. Conservative management was determined as the use of antibiotics only (i.e. an intervention was not offered at initial consultation). Interventional radiology (IR) guided drain insertion refers to CT or ultrasound (US) guided insertion of an intra-abdominal drain. Time to theatre was calculated in hours from the admission time to the start of the operation. Operative time was calculated in minutes from skin incision to the end of skin closure. Time of day when the procedure was performed was determined by the start time of the operation, with those starting after 17:00 until the following day at 08:00 classified to have been performed out of hours.

Operative details were recorded based on the operating surgeon's documentation. Conversion from a laparoscopic to open approach was determined as additional incisions performed either in the right iliac fossa or midline laparotomy. The level of the surgeon was determined based on the years of practice post-qualification (Junior Trainee; Senior Trainee; Consultant). Critical care admission was determined if the patient was cared for in a Level 2 (high dependency unit) or a Level 3 care (intensive care unit) setting. Re-attendance referred to any patient re-presenting following their initial admission. This study has been reported in line with the STROCSS criteria (14).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years old and above
* Confirmed diagnosis of acute appendicitis

Exclusion Criteria:

* Patients aged less than 16 years old

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in this study were all adults (≥16 years) with a diagnosis of acute appendicitis made clinically and/or radiologically in our hospital. Patients presented sequentially to the emergency department, and subsequently were referred to the emergency surgical service for further management.
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-05 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Mortality | within 90 days of a patient's initial presentation
  Death secondary to acute appendicitis
Failure of primary proposed treatment | within 90 days of a patient's initial presentation
  failure of conservative management and need to undergo surgery

SECONDARY OUTCOMES:
length of stay | within 90 days of a patient's initial presentation
  length of stay in hospital from admission date till discharge date or death
Re-attendance | within 90 days of a patient's initial presentation
  Re-attendance to hospital after patient's discharge whether planned or unplanned
Imaging | within 90 days of a patient's initial presentation
  imaging modality obtained and findings to confirm the diagnosis of acute appendicitis
Intra-operative findings during surgery | within 90 days of a patient's initial presentation
  Intra-operative findings of pus or free fluid during appendicectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrooke's University Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As individual participant data contain private confidential data, this data will not be shared or made available publicly however the primary would be to answer or clarify any relevant queries.